CLINICAL TRIAL: NCT04230330
Title: A Pilot Study of Nivolumab in Combination With GDP (Gemcitabine, Dexamethasone, Cisplatin)/ L-asparaginase in Patients With Advanced Stage or Relapsed/ Refractory Natural-killer/ T-cell Lymphoma
Brief Title: Nivolumab in Combination With GDP/ L-asparaginase in NK/ T-cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI has left the institution.
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-8R6
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: NK/T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Nivolumab; Gemcitabine; Cisplatin; Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental): After 4 doses of nivolumab, if the patient has complete responses (CR) or good partial response (PR), the patient will continue on nivolumab until disease progression, unacceptable toxicities, or discontinuation of treatment. During PET4-directed treatment with single agent nivolumab, if patient has PD, they will proceed to the Nivo+GDP/L-aspa arm.
  Interventions: Drug: IV Nivolumab
- Nivolumab + GDP/ L-asparaginase (Experimental): After 4 doses of nivolumab, if the patient has PR, stable disease (SD), or progressive disease (PD), the patient will switch to nivolumab-GDP/L-aspa treatment. After 6 cycles of treatment, if CR is achieved, the patient will continue on single agent nivolumab until disease progression, unacceptable toxicities, or discontinuation of treatment.
  Interventions: Drug: IV Nivolumab; Drug: IV Gemcitabine; Drug: IV Cisplatin; Drug: IV/PO Dexamethasone; Drug: IV L-asparaginase

INTERVENTIONS:
Drug: IV Nivolumab — 240mg every 2 weeks.
  Other Names: Opdivo
  Arms: Nivolumab
Drug: IV Nivolumab — Initial treatment dose is 240mg every 2 weeks for 4 doses. Dose changes to 360mg every 3 weeks when given with GDP/L-aspa. Maintenance treatment dose is 240mg every 2 weeks.
  Other Names: Opdivo
  Arms: Nivolumab + GDP/ L-asparaginase
Drug: IV Gemcitabine — 800mg/m2 on Days 1 and 8 every 21 days
  Arms: Nivolumab + GDP/ L-asparaginase
Drug: IV Cisplatin — 20mg/m2 on Day 1 to 4 every 21 days
  Arms: Nivolumab + GDP/ L-asparaginase
Drug: IV/PO Dexamethasone — 10mg on Days 1 to 4 every 21 days
  Arms: Nivolumab + GDP/ L-asparaginase
Drug: IV L-asparaginase — 6000 Units/m2 on Days 2 to 8 every 21 days
  Arms: Nivolumab + GDP/ L-asparaginase

SUMMARY:
This is a pilot study investigating the role of nivolumab, a PD-1 inhibitor, in the treatment of advanced stage or relapsed/refractory NKTL. Patients who have received PD-1 inhibitors will be excluded from this study.

Patients who have a complete response or good partial response to nivolumab during initial phase will continue to be treated with nivolumab. Patients who have a partial response, stable disease, and progressive disease to nivolumab during initial phase will be treated with the combination of nivolumab and GDP/L-asparaginase.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent

  * Subjects must have signed and dated and IRB-approved written consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal subject care
  * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study
* Target population

  * All subjects must have histologically confirmed extranodal natural-killer/T-cell lymphoma (NKTL)
  * Subjects must have

    * previously untreated stage III or IV NKTL, OR
    * relapsed/refractory NKTL who has received at least 2 cycles of one prior regimen or previous radiotherapy administered with curative intent and one of the following:

      * Failed to achieve at least a partial response
      * Failed to achieve a complete response at the end of planned therapy with curative intent
      * Progressed after initial response
  * Age ≥ 21 years
  * ECOG Performance status 0 - 2
  * Subjects must have laboratory test results within these ranges:

    * Absolute neutrophil count (ANC) ≥ 1.5 x10^9/L
    * Platelet count ≥ 75 x10^9/L
    * Creatinine clearance ≥ 40ml/min
    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN). Higher levels are acceptable if these can be attributed to active haemolysis or ineffective erythropoiesis
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2x ULN
* Women of childbearing potential (WOCBT) must agree to use dual methods of contraception and have a negative serum or urine pregnancy test prior study treatment. Male patients must use an effective barrier method of contraception if sexually active with a WOCBT

Exclusion Criteria:

* Previous treatment with an anti PD-1, anti PD-L1, anti PD-L2, anti-CD137, or anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Previous GDP therapy
* Previous serious hypersensitivity reaction or symptomatic pancreatitis from L-asparaginase
* Uncontrolled central nervous (CNS) disease
* Uncontrolled hepatitis B or C
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (NCI CTCAE version 4) or baseline before administration of study drug
* Subjects with > grade 1 peripheral neuropathy
* Any serious or uncontrolled medical disorder, autoimmune disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration or would impair the ability fo the subject to receive the study drug
* Subjects who have had prior malignancies (other than NKTL) for ≤5 year with exception of currently treated basal cell, squamous cell carcinoma of the skin or carcinoma "in situ" of the cervix or breast.
* Subjects who have had other anti-cancer therapy including radiation or experimental drug therapy within 28 days of enrollment
* Subjects with known allergies or hypersensitivities to the study drugs
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
* Pregnant women or women who are breastfeeding are excluded from this study

Inclusion of women and minorities:

Men and women of all ethnic groups are eligible for this study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete response and partial response to treatment | 6 months after the start of treatment
  To calculate best overall response rate
Number of incidences of grade 3-5 non-haematological adverse events | From start of first treatment to 100 days after last treatment dose
  To calculate the toxicity rate of the treatment

SECONDARY OUTCOMES:
Progression-free survival | From start of treatment to date of disease progression or death, up to 2.5 years
Overall survival | From the start of treatment to date of death from any cause, up to 2.5 years
Number of patients with complete response and partial response to single agent nivolumab | 6 months after the start of treatment
  To calculate the overall response rate of single agent nivolumab
Number of patients with complete response and partial response to nivolumab in combination with GDP/L-asparaginase | 6 months after the start of treatment
Number of incidences of adverse events | From start of first treatment to 100 days after last treatment dose
  To calculate the rate of adverse events from nivolumab with or without GDP/L-asparaginase

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Tang, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

REFERENCES:
- [Background] Li X, Cheng Y, Zhang M, Yan J, Li L, Fu X, Zhang X, Chang Y, Sun Z, Yu H, Zhang L, Wang X, Wu J, Li Z, Nan F, Tian L, Li W, Young KH. Activity of pembrolizumab in relapsed/refractory NK/T-cell lymphoma. J Hematol Oncol. 2018 Jan 31;11(1):15. doi: 10.1186/s13045-018-0559-7. PMID 29386072
- [Background] Kwong YL, Chan TSY, Tan D, Kim SJ, Poon LM, Mow B, Khong PL, Loong F, Au-Yeung R, Iqbal J, Phipps C, Tse E. PD1 blockade with pembrolizumab is highly effective in relapsed or refractory NK/T-cell lymphoma failing l-asparaginase. Blood. 2017 Apr 27;129(17):2437-2442. doi: 10.1182/blood-2016-12-756841. Epub 2017 Feb 10. PMID 28188133